CLINICAL TRIAL: NCT03265522
Title: The Development and Pilot Testing of Tailored Mediterranean Lifestyle Education to Encourage Behaviour Change in Patients With Mild Cognitive Impairment
Brief Title: Tailored Mediterranean Lifestyle Education in Patients With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Principal Investigator, Jayne Woodside, PhD, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16/NI/0105
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Mild Cognitive Impairment
Keywords: Mediterranean diet; Lifestyle
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: "ThinkMed" resource at baseline (Experimental): The "ThinkMed" resource contains an information booklet, recipe books, menu plan cards, shopping list cards and goal setting cards. Participants will receive this resource on one occasion at baseline (n=20)
  Interventions: Behavioral: "ThinkMed" resource at baseline
- Group 2: "ThinkMed" resource (staged) (Experimental): This group of participants will receive the "ThinkMed" resource at monthly intervals for 5 months accompanied by telephone feedback from the research dietitian (n=20)
  Interventions: Behavioral: "ThinkMed" resource (staged)
- Group 3: Standard Care (control) group (Placebo Comparator): Participants will continue with the standard care provided by their physician. Participants will receive the "ThinkMed" resource after their final 6 month study visit (i.e. delayed intervention) (n=20)
  Interventions: Behavioral: Standard Care Control

INTERVENTIONS:
Behavioral: "ThinkMed" resource at baseline — The "ThinkMed" resource contains an information booklet, recipe books, menu plan cards, shopping list cards and goal setting cards. Participants will receive this resource on one occasion at baseline.
  Arms: Group 1: "ThinkMed" resource at baseline
Behavioral: Standard Care Control — Participants will continue with the standard care provided by their physician. Participants will receive the "ThinkMed" resource after their final 6 month study visit (i.e. delayed intervention).
  Arms: Group 3: Standard Care (control) group
Behavioral: "ThinkMed" resource (staged) — This group of participants will receive the "ThinkMed" resource at monthly intervals for 5 months accompanied by telephone feedback from the research dietitian
  Arms: Group 2: "ThinkMed" resource (staged)

SUMMARY:
Evidence suggests that a Mediterranean diet can have a beneficial effect on brain health. Mild cognitive impairment (MCI) describes problems with brain function such as difficulty with day-to-day memory and concentration. It is at this stage that Mediterranean diet could prove beneficial in terms of prevention.

Previous research by Queens University investigated the opinions of patients with MCI and their care givers to inform the development of Mediterranean diet education material to encourage behaviour change. The study suggested that MCI patients lacked awareness of the link between Mediterranean diet and brain function, although were interested to learn more. Feedback on the developed educational material was positive although there were suggested improvements such as tailoring information to memory loss, a potential staged approach to delivery and adaptations to the material content.

This present study aims to pilot test refined educational material among MCI participants to evaluate the feasibility of encouraging dietary behaviour change among this patient group.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility of a theory-based, tailored Mediterranean lifestyle education intervention to encourage behaviour change in patients with MCI. The proposed study will be a 6 month RCT with a total of 60 MCI patients who will be randomised to 1 of 3 groups:

1. Group 1 will receive the Mediterranean lifestyle education resource on one occasion at baseline
2. Group 2 will receive the Mediterranean lifestyle education resource at monthly intervals for 5 months accompanied by telephone feedback from the research dietitian
3. Group 3 will receive standard care (control group). Participants will receive the Mediterranean lifestyle education resource after their final 6 month study visit (i.e. delayed intervention).

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Mild Cognitive Impairment by their physician
* Mediterranean diet score (MDS) less than or equal to 4 (Estruch et al., 2006)
* Willing to make changes to their diet

Exclusion Criteria:

* Diagnosis of dementia
* Patients with visual or English language impairment
* Psychiatric problems
* Significant medical comorbidity
* Body Mass Index (BMI) ≤ 19 and ≥ 40 kg/m2
* Excessive alcohol consumption
* Taking high dose nutritional supplements
* Dietary restrictions/allergies that would substantially limit ability to complete study requirements
* Inability to provide informed consent
* History of, or comorbid condition which may alter performance on cognitive tests e.g. stroke, head injury, Parkinson's disease, learning disability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Mediterranean Diet Score (MDS) at 6 months | Baseline, 6 months
  Mediterranean dietary intake will be measured by a validated questionnaire

SECONDARY OUTCOMES:
Physical Activity | Baseline, 6 months
  RPAQ-Recent Physical Activity Questionnaire
Anthropometric measurements | Baseline, 6 months
  Weight and height measurements to calculate BMI
Muscle Strength | Baseline, 6 months
  Measured using a grip-strength dynamometer
Geriatric Depression Scale | Baseline, 6 months
  Geriatric Depression Scale Questionnaire
Functional Assessment (1) | Baseline, 6 months
  Measured by the instrumental activities of daily living scale (IADL) by Lawton and Brody (1969) questionnaire
Cognitive Assessment | Baseline, 6 months
  A comprehensive cognitive assessment will be performed, including: global cognition, motor skills, executive function episodic/visual memory, and information processing and sustained attention using a validated neuropsychological test battery (Cantab Cognitive Battery, Cambridge Cognition Ltd.)
Barriers to consuming a Mediterranean Diet questionnaire | Baseline, 6 months
  Dietary behaviour change questionnaire to measure adherence to a Mediterranean diet
Blood Sample | Baseline, 6 months
  A blood sample will be taken from participants to be stored for analysis of biomarkers of MD adherence and biomarkers of neurodegenerative disease risk.
Functional Assessment (2) | Baseline, 6 months
  Measured by the Bristol activities of daily living scale (Bucks et al. 1996) questionnaire
4-day Food Diary | Baseline, 6 months
  A food diary will be completed to assess compliance with a Mediterranean diet
Change in Lifestyle questionnaire | Baseline, 6 months
  A questionnaire to measure change in lifestyle behaviours
Dietary Quality of Life questionnaire | Baseline, 6 months
  A questionnaire to measure dietary quality of life
Mediterranean Diet Knowledge questionnaire | Baseline, 6 months
  A questionnaire to measure participants Mediterranean diet knowledge
Rand SF-36 HEALTH SURVEY | Baseline, 6 months
  A questionnaire to measure participants views and beliefs on health
Staging Algorithm Questionnaire | Baseline, 6 months
  A questionnaire to measure participants readiness to change their diet and lifestyle
Mediterranean Diet self-efficacy questionnaire | Baseline, 6 months
  A questionnaire to measure participants self-efficacy
Mediterranean diet tolerance questionnaire | Baseline, 6 months
  A questionnaire to measure tolerance to a Mediterranean diet

OTHER OUTCOMES:
Process Evaluation (1) - telephone contact evaluation | up to 3 months post intervention
  Determination individual participation and engagement with the intervention by reviewing telephone contact log record and telephone checklist evaluation
Process Evaluation (2) - study records | up to 3 months post intervention
  A review of study records- including attrition rates, reason for dropout
Process Evaluation (3) - structured interviews | up to 3 months post intervention
  Post intervention structured interviews for participant evaluation of the intervention programme and dietary educational materials

CONTACTS AND LOCATIONS:
Overall Officials: Jayne Woodside, PhD, Principal Investigator — Queens University Belfast
Locations (1):
- Belfast Health and Social Care Trust, Belfast, United Kingdom

REFERENCES:
- [Derived] McGrattan AM, McEvoy CT, Vijayakumar A, Moore SE, Neville CE, McGuinness B, McKinley MC, Woodside JV. A mixed methods pilot randomised controlled trial to develop and evaluate the feasibility of a Mediterranean diet and lifestyle education intervention 'THINK-MED' among people with cognitive impairment. Pilot Feasibility Stud. 2021 Jan 4;7(1):3. doi: 10.1186/s40814-020-00738-3. PMID 33390187